CLINICAL TRIAL: NCT05502250
Title: Tislelizumab Plus Gemcitabine and Cisplatin for Relapsed or Refractory Hodgkin Lymphoma Followed by Tislelizumab Consolidation in Patients in Metabolic Complete Remission (TIGERR-HL). An Open Label Phase II Trial
Brief Title: Tislelizumab, Gemcitabine and Cisplatin for R/R Hodgkin Lymphoma Followed by Tislelizumab Consolidation in Patients in Metabolic Complete Remission
Acronym: HOVON164HL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Stichting Hemato-Oncologie voor Volwassenen Nederland (Other)
Collaborators: Danish Lymphoma Group (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HO164; 2022-502225-17 (Other: EMA Clinical Trials Information System (CTIS))
Record Dates: First submitted 2022-05-25; First posted 2022-08-16 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Hodgkin Lymphoma
MeSH Terms: conditions — Hodgkin Disease | interventions — Gemcitabine; Cisplatin; tislelizumab

STUDY DESIGN:
Intervention Model Description: Single arm = 4 cycles of gemcitabine and cisplatin (GP) + tislelizumab followed by 13 cycles of tislelizumab
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single-arm (Experimental): 4 cycles of gemcitabine and cisplatin (GP) + tislelizumab followed by 13 cycles of tislelizumab
  Interventions: Drug: gemcitabine, cisplatin and tislelizumab

INTERVENTIONS:
Drug: gemcitabine, cisplatin and tislelizumab — All patients will receive 2 cycles of gemcitabine and cisplatin (GP) + tislelizumab. Each cycle lasts 21 days. Treatment is given through an IV line on day 1 and 8.
  After 2 cycles a FDG-PET-CT scan will be performed. Patients who respond well will proceed with 2 additional cycles of GP + tislelizumab . Patients with insufficient response will stop with the study treatment and they will continue treatment according to local practice.
  After 4 cycles of GP + tislelizumab another FDG-PET-CT scan will be performed. If this scan shows that the disease is under control (metabolic complete remission) patients will proceed with 13 cycles of tislelizumab consolidation treatment (21 day cycles). Treatment is given on day 1 through an IV line.

SUMMARY:
This trial investigates the efficacy and safety of the drug tislelizumab in combination with chemotherapy as a treatment for patients with R/R HL. Tislelizumab is given in combination with chemotherapy (gemcitabine and cisplatin) followed by consolidation with tislelizumab alone. The study primary question is whether this strategy works as well as the standard treatment with intensive chemotherapy and autologous stem cell transplant.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed classical HL (according to the latest version of the WHO classification).
* Primary refractory to first line chemotherapy, or in first relapse after any polychemotherapy regimen (e.g. ABVD, baseline BEACOPP or escalated BEACOPP, or other induction regimens).
* In case of relapse, the relapse must be histologically confirmed. In case histologic biopsy is not possible, at least confirmation of the relapse by fine needle aspirate (FNA) or sequential imaging is required.
* Measurable disease, based on Lugano criteria 2014 [40]; i.e. CT scans showing at least 2 or more clearly demarcated lesions with a long axis ≥ 1.5 cm and a short axis diameter ≥ 1.0 cm, or 1 clearly demarcated lesion with a long axis ≥ 2.0 cm and a short axis diameter ≥ 1.0 cm. These lesions must be FDG-PET-positive.
* Age 18-70 years inclusive.
* WHO/ECOG Performance Status ≤ 1 (see appendix C).
* No major organ dysfunction, unless HL-related:

  * Total bilirubin < 1.5x ULN (unless due to lymphoma involvement of the liver or a known history of Gilbert's syndrome; in that case bilirubin may be elevated up to 3 x ULN).
  * ALT/AST < 3x ULN (unless due to lymphoma involvement of the liver; in that case ALT/AST may be elevated up to 5 x ULN).
  * GFR > 60 ml/min as estimated by the Cockcroft&Gault formula.
* Adequate BM function defined as:

  * Absolute neutrophil count ≥ 1.5x109/L, unless caused by diffuse bone marrow infiltration by the HL.
  * Platelets ≥ 75 x109/L, unless caused by diffuse bone marrow infiltration by the HL.
  * Hemoglobin must be ≥ 8 g/dL (5 mmol/L).
* Resolution of toxicities from first-line therapy.
* Able to adhere to the study visit schedule and other protocol requirements.
* Negative pregnancy test at study entry.
* Female patient is either post-menopausal for at least 1 year before the screening visit or surgically sterile or if of childbearing potential, agrees to practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent through at least 6 months after the last dose of study drug, or agrees to completely abstain from heterosexual intercourse.
* Male patient, even if surgically sterilized, (i.e., status post vasectomy) agrees to practice effective barrier contraception during the entire study period and through 6 months after the last dose of study drug, or agrees to completely abstain from heterosexual intercourse.
* Written informed consent.
* Patient is capable of giving informed consent.

Exclusion Criteria:

* Previous treatment with an PD-1 or PDL-1 blocking agent.
* Patients who have been using other investigational agents within at least 5 half lives or 4 weeks, whichever is longer, of the most recent agent used prior to start of protocol treatment.
* Patients who were treated with myelosuppressive chemotherapy or biological therapy within at least 5 half lives or 4 weeks, whichever is longer, before start of protocol treatment.
* Patients who were treated with steroids for more than 25 mg /day for at least 14 days before start of protocol treatment.
* Patients receiving radiation therapy within 2 weeks prior to start of protocol treatment. Emergency radiation therapy is allowed, as long as measurable disease (at non-irradiated sites) persists.
* Prior allogeneic stem cell transplantation or solid organ transplantation.
* Peripheral neuropathy > grade 2.
* Active autoimmune diseases or history of autoimmune diseases that may relapse.

Note: Patients with the following diseases are not excluded and may proceed to further screening:

* Controlled Type I diabetes.
* Hypothyroidism (provided it is managed with hormone replacement therapy only).
* Controlled celiac disease.
* Skin diseases not requiring systemic treatment (eg, vitiligo, psoriasis, alopecia).
* Any other auto-immune disease that is not expected to recur due to the protocol treatment.

  * Any condition that required systemic treatment with either corticosteroids (> 10 mg daily of prednisone or equivalent) or other immunosuppressive medication ≤ 14 days before study treatment.

Note: Patients who are currently or have previously been on any of the following steroid regimens are not excluded:

* Adrenal replacement steroid (dose ≤ 10 mg daily of prednisone or equivalent).
* Topical, ocular, intra-articular, intranasal, or inhaled corticosteroid with minimal systemic absorption.
* Short course (≤ 7 days) of corticosteroid prescribed prophylactically (eg, for contrast dye allergy) or for the treatment of a non-autoimmune condition (eg, delayed-type hypersensitivity reaction caused by contact allergen).

  * History of interstitial lung disease, non-infectious pneumonitis or uncontrolled diseases including pulmonary fibrosis, acute lung diseases, etc.
  * Known cerebral or meningeal disease (HL or any other etiology), including signs or symptoms of progressive multifocal leukoencephalopathy (PML).
  * Patients who have a history of another primary malignancy less than 2 years before study inclusion or previously diagnosed with another malignancy and have evidence of residual disease, with the exception of non-melanoma skin cancer, completely resected melanoma TNMpT1 and carcinoma in situ of the uterine cervix.
  * Patients with any active systemic viral, bacterial, or fungal infection requiring systemic antibiotics within 2 weeks prior to first study drug dose.
  * Patients with active HIV (unless viral load undetectable and CD4 counts within the normal range under antiretroviral therapy), active HBV (e.g. HBV DNA PCR positive or HBV surface antigen-positivity), or active HCV (e.g. HCV RNA detected). Patients with inactive HBV are eligible, but antiviral prophylaxis is obligatory.
  * Patients who have any severe and/or uncontrolled cardiovascular condition that could affect their participation in the study such as:
* Known history of symptomatic congestive heart failure (NYHA III, IV), myocardial infarction ≤ 6 months prior to first study drug.
* Evidence of current serious uncontrolled cardiac arrhythmia, angina pectoris, electrocardiographic evidence of acute ischemia or active conduction system abnormalities.
* History of cerebrovascular accident ≤ 6 months before study treatment.

  * Patient who was administered a live vaccine ≤ 4 weeks before study treatment.
  * A history of severe hypersensitivity reactions to chimeric or humanized antibodies or platinum-based compounds.
  * Breast-feeding female patients.
  * Current participation in another clinical trial with medicinal products.
  * Any psychological, familial, sociological and geographical condition potentially hampering compliance with the study protocol and follow-up schedule.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2023-07-14 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2030-04 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) probability at 2 years after registration. PFS is defined as time from registration to progression or death from any cause, whichever comes first. | Approximately up to 48 months following first patient enrollment
  Single-arm

SECONDARY OUTCOMES:
Overall response rate (ORR: mCR and mPR rates) (as assessed by FDG-PET/CT) after 2 and 4 cycles of tislelizumab in combination with GP chemotherapy induction. | Approximately up to 28 months following first patient enrollment
  Single-arm
Rate of CTCAE grade 3/4 toxicities of tislelizumab in combination with GP chemotherapy. | Approximately up to 28 months following first patient enrollment
  Single-arm
Rate of CTCAE grade 2 to 4 immune related toxicities of tislelizumab in combination with GP chemotherapy. | Approximately up to 36 months following first patient enrollment
  Single-arm
Rate of CTCAE grade 3/4 toxicities of tislelizumab consolidation treatment. | Approximately up to 36 months following first patient enrollment
  Single-arm
Progression free survival (PFS) as time-to-event outcome. | Approximately up to 36 months following first patient enrollment
  Single-arm
Event free survival (EFS) defined as time from registration to start new HL treatment, progression or death from any cause, whichever comes first. | Approximately up to 84 months following first patient enrollment
  Single-arm
Disease free survival (DFS) defined as time from start of consolidation therapy to relapse or death from any cause, whichever comes first. | Approximately up to 84 months following first patient enrollment
  Single-arm
Overall survival (OS) defined as time from registration to death from any cause. | Approximately up to 84 months following first patient enrollment
  Single-arm

CONTACTS AND LOCATIONS:
Locations (15):
- BE-Bruxelles-STLUC, Brussels, Belgium
- Denmark (3):
  - DK-Aarhus N-AUH, Aarhus
  - DK-Copenhagen-RIGSHOSPITALET, Copenhagen
  - DK-Odense-OUH, Odense
- Netherlands (11):
  - NL-Amersfoort-MEANDERMC, Amersfoort
  - NL-Amsterdam-AMC, Amsterdam
  - NL-Arnhem-RIJNSTATE, Arnhem
  - NL-Eindhoven-MAXIMAMC, Eindhoven
  - NL-Goes-ADRZ, Goes
  - NL-Groningen-UMCG, Groningen
  - NL-Hoofddorp-SPAARNEGASTHUIS, Hoofddorp
  - NL-Leeuwarden-MCL, Leeuwarden
  - NL-Maastricht-MUMC, Maastricht
  - NL-Rotterdam-ERASMUSMC, Rotterdam
  - NL-Den Haag-HAGA, The Hague

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Website of HOVON - the Haemato Oncology Foundation for Adults in the Netherlands — https://hovon.nl/en